CLINICAL TRIAL: NCT05796245
Title: Infliximab-Pfizer Biosimilar Post-Marketing Database Study
Brief Title: A Study to Learn About the Study Medicine Called Infliximab (Genetical Recombination)[Infliximab Biosimilar 3] in People With Rheumatoid Arthritis, Ulcerative Colitis, Crohn's Disease, or Psoriasis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B5371010; NCT05796245 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-03-02; First posted 2023-04-03 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Arthritis, Rheumatoid; Colitis, Ulcerative; Crohn Disease; Psoriasis
Keywords: Tumor Necrosis Factor, TNF; Infliximab; Biosimilar
MeSH Terms: conditions — Arthritis, Rheumatoid; Colitis, Ulcerative; Crohn Disease; Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infliximab (Genetical Recombination)[Infliximab Biosimilar 3]
- Remicade

SUMMARY:
The purpose of this study is to learn about the safety of the safety of the study medicine called infliximab for the possible treatment of rheumatoid arthritis (RA), ulcerative colitis (UC, Crohn's disease, or psoriasis.

RA is a kind of joint disease that causes pain and swelling.

UC causes inflammation and sores (also called ulcers), in the lining of the rectum and colon.

Chron's disease is a disease that lasts for a long time and causes severe irritation in your digestive tract.

Psoriasis is a skin disease that gives you a dry, scaly rash.

The study includes patient's data from the database who:

* Have at least 90 days of look-back period
* Have any of these diseases (RA, UC, Crohn's disease, or Psoriasis) in the 90-day look back period
* Are 15 years of age or older at the time of first dosing

All the patient's data included in this study would have received infliximab as intravenous (into veins) injection.

ELIGIBILITY:
Inclusion criteria

1. Have at least 90 days of look-back period
2. Have diagnostic code of indicated diseases (rheumatoid arthritis, ulcerative colitis, Crohn's disease, or psoriasis) in the 90-day look-back period. Patients with >1 indication will be summarized as a separate group from each sub-cohort. An inpatient or outpatient visit assigned a diagnosis code consistent with either rheumatoid arthritis, ulcerative colitis, Crohn's disease, or psoriasis using ICD-10 coding.
3. 15 years of age or older at the time of index date

Exclusion criteria

1. Patients with pre-existing safety outcome event during the 90-day look-back period will be excluded from the study cohort for that specific outcome event as this study is observing incident cases.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes individuals who have a diagnosis of rheumatoid arthritis, ulcerative colitis, Crohn's disease, or psoriasis and have been exposed to Infliximab-Pfizer Biosimilar or the innovator (Remicade) with a planned study period between December 1, 2018 and November 30, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 2207 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B5371010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of study patients were extracted from the Medical Data Vision (MDV) database according to the study entry criteria. MDV database is a hospital-based claims database in Japan that consists of outpatient and inpatient data from hospitals using the diagnosis procedure combination system. The study period was from December 1, 2018 through November 30, 2023.
Groups:
- Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3]: Patients treated with Infliximab-Pfizer Biosimilar who meet the inclusion/exclusion criteria.
- Remicade (Infliximab [Genetical Recombination]): Patients treated with Remicade who meet the inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] | Remicade (Infliximab [Genetical Recombination])
Started (Main cohort) | 92 | 2115
Full Analysis Set (Patients who were diagnosed with rheumatoid arthritis, ulcerative colitis, or Crohn's disease; received Infliximab-Pfizer Biosimilar or Remicade; were aged 15 years or older at the index date; and had at least 90 days of look-back period. Patients with pre-existing safety outcome event during the 90-day look-back period were excluded from the study cohort of the respective outcome event.) | 92 | 2115
Comparative Analysis Set (Patients who received Infliximab-Pfizer Biosimilar and Remicade. The comparative analysis set was a subset of the full analysis set who were new users. That is, patients switching from non-Pfizer Infliximab Biosimilar or Remicade to Infliximab-Pfizer Biosimilar were excluded. Also, patients switching from any Infliximab Biosimilar to Remicade were excluded.) | 28 | 2115
Completed | 92 | 2115
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of the patients who were main cohort in the study, those who met the eligibility criteria were included in the following analysis sets: Full analysis set (Infliximab-Pfizer Biosimilar), n=92; Full analysis set (Remicade), n=2115; Comparative analysis set (Infliximab-Pfizer Biosimilar), n=28; and Comparative analysis set (Remicade), n=2115.
Groups:
- Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] (Full Analysis Set): Patients treated with Infliximab-Pfizer Biosimilar who meet the inclusion/exclusion criteria.
- Remicade (Infliximab [Genetical Recombination]) (Full Analysis Set): Patients treated with Remicade who meet the inclusion/exclusion criteria.
- Total: Total of all reporting groups
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] (Full Analysis Set) | Remicade (Infliximab [Genetical Recombination]) (Full Analysis Set) | Total
Number analyzed (Participants) | 92 | 2115 | 2207
Age, Customized [Number; unit: Participants] — Population: The full analysis set included all patients who were considered eligible by the inclusion and exclusion criteria. The comparative analysis set was a subset of the full analysis set who were new users.
  Participants
    <18 years (Full analysis set) | 1 | 88 | 89
    ≥18 and <65 years (Full analysis set) | 52 | 1615 | 1667
    ≥65 years (Full analysis set) | 39 | 412 | 451
    <18 years (Comparative analysis set): number analyzed (Participants) | 28 | 2115 | 2143
    <18 years (Comparative analysis set) | 1 | 88 | 89
    ≥18 and <65 years (Comparative analysis set): number analyzed (Participants) | 28 | 2115 | 2143
    ≥18 and <65 years (Comparative analysis set) | 18 | 1615 | 1633
    ≥65 years (Comparative analysis set): number analyzed (Participants) | 28 | 2115 | 2143
    ≥65 years (Comparative analysis set) | 9 | 412 | 421
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The full analysis set included all patients who were considered eligible by the inclusion and exclusion criteria. The comparative analysis set was a subset of the full analysis set who were new users.
  Participants
    Full analysis set: Female | 49 | 827 | 876
    Full analysis set: Male | 43 | 1288 | 1331
    Comparative analysis set: number analyzed (Participants) | 28 | 2115 | 2143
    Comparative analysis set: Female | 17 | 827 | 844
    Comparative analysis set: Male | 11 | 1288 | 1299
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Serious Infections
Description: The observation of serious infections was expected to occur in an acute time period following any exposure. An incident event occurring during the 60-day risk window was counted in the numerator for the analysis and the person-time accrued until the first occurrence of an event, the end of the 60-day risk window, date of switch treatment, death, or the end of study period. Additionally, two types of analyses based on propensity score were conducted.
  For the full analysis set, 9 and 232 events occurred with a total of 151.9 and 2609.9 person-years in the Infliximab-Pfizer Biosimilar group and Remicade group, respectively. For the comparative analysis set, 5 and 232 events occurred with a total of 22.8 and 2609.9 person-years. For the comparative analysis set (IPTW weighted), 0.5 and 230.7 events occurred with a total of 3.6 and 2598.5 person-years. For the comparative matched analysis set, 5 and 6 events occurred with a total of 22.8 and 46.7 person-years.
Time Frame: From index date up to 60 days after last dose
Population: For the analysis of each outcome event, those patients experiencing the same outcome event during the 90-day look-back period prior to the index date were excluded. For serious infections, this resulted in Full analysis set (Infliximab-Pfizer Biosimilar, n=86; Remicade, n=1909), Comparative analysis set (Infliximab-Pfizer Biosimilar, n=23; Remicade, n=1909).
Measure: Number; unit: serious infections per 1 person-year
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] | Remicade (Infliximab [Genetical Recombination])
Number analyzed (Participants) | 92 | 2115
serious infections per 1 person-year
  Incidence rate of serious infections (Full analysis set): number analyzed (Participants) | 86 | 1909
  Incidence rate of serious infections (Full analysis set) | 0.06 | 0.09
  Incidence rate of serious infections (Comparative analysis set): number analyzed (Participants) | 23 | 1909
  Incidence rate of serious infections (Comparative analysis set) | 0.22 | 0.09
  Incidence rate of serious infections (Comparative analysis set, IPTW weighted): number analyzed (Participants) | 23 | 1909
  Incidence rate of serious infections (Comparative analysis set, IPTW weighted) | 0.13 | 0.09
  Incidence rate of serious infections (Comparative matched analysis set): number analyzed (Participants) | 23 | 46
  Incidence rate of serious infections (Comparative matched analysis set) | 0.22 | 0.13
Statistical Analysis 1: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set, IPTW weighted; Test type: Other — Estimation; Cox Proportional Hazard = 1.43, 95% CI 2-sided [0.39 to 5.20] — Hazard Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 2: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set, IPTW weighted; Test type: Other — Estimation; Risk Ratio (RR) = 1.43, 95% CI 2-sided [0.38 to 5.34] — Risk Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 3: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set, IPTW weighted; Test type: Other — Estimation; Risk Difference (RD) = 0.04, 95% CI 2-sided [-0.20 to 0.11] — Risk Difference (Exposed-Reference), where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 4: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative matched analysis set; Test type: Other — Estimation; Cox Proportional Hazard = 1.63, 95% CI 2-sided [0.54 to 4.90] — Hazard Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 5: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative matched analysis set; Test type: Other — Estimation; Risk Ratio (RR) = 1.71, 95% CI 2-sided [0.55 to 5.26] — Risk Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 6: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative matched analysis set; Test type: Other — Estimation; Risk Difference (RD) = 0.09, 95% CI 2-sided [-0.10 to 0.39] — Risk Difference (Exposed-Reference), where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 7: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set; Test type: Other — Estimation; Cox Proportional Hazard = 2.44, 95% CI 2-sided [1.05 to 5.67] — Crude Hazard Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 8: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set; Test type: Other — Estimation; Risk Ratio (RR) = 2.47, 95% CI 2-sided [1.02 to 5.99] — Crude Risk Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 9: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set; Test type: Other — Estimation; Risk Difference (RD) = 0.13, 95% CI 2-sided [-0.06 to 0.32] — Crude Risk Difference (Exposed-Reference), where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade

2. Secondary Outcome: Incidence Rate of Tuberculosis
Description: The observation of tuberculosis was expected to occur in an acute time period following any exposure. An incident event occurring during the 60-day risk window was counted in the numerator for the analysis and the person-time accrued until the first occurrence of an event, the end of the 60-day risk window, date of switch treatment, death, or the end of study period. Additionally, two types of analyses based on propensity score were conducted.
  For the full analysis set, 0 and 14 events occurred with a total of 161.8 and 2904.1 person-years in the Infliximab-Pfizer Biosimilar group and Remicade group, respectively. For the comparative analysis set, 0 and 14 events occurred with a total of 27.2 and 2904.1 person-years. For the comparative analysis set (IPTW weighted), 0.0 and 14.3 events occurred with a total of 10.4 and 2889.7 person-years. For the comparative matched analysis set, 0 and 1 event occurred with a total of 27.2 and 50.1 person-years.
Time Frame: From index date up to 60 days after last dose
Population: For the analysis of each outcome event, those patients experiencing the same outcome event during the 90-day look-back period prior to the index date were excluded. For tuberculosis, this resulted in Full analysis set (Infliximab-Pfizer Biosimilar, n=91; Remicade, n=2100), Comparative analysis set (Infliximab-Pfizer Biosimilar, n=28; Remicade, n=2100).
Measure: Number; unit: tuberculosis per 1 person-year
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] | Remicade (Infliximab [Genetical Recombination])
Number analyzed (Participants) | 92 | 2115
tuberculosis per 1 person-year
  Incidence rate of tuberculosis (Full analysis set): number analyzed (Participants) | 91 | 2100
  Incidence rate of tuberculosis (Full analysis set) | 0.00 | 0.00
  Incidence rate of tuberculosis (Comparative analysis set): number analyzed (Participants) | 28 | 2100
  Incidence rate of tuberculosis (Comparative analysis set) | 0.00 | 0.00
  Incidence rate of tuberculosis (Comparative analysis set, IPTW weighted): number analyzed (Participants) | 28 | 2100
  Incidence rate of tuberculosis (Comparative analysis set, IPTW weighted) | 0.00 | 0.00
  Incidence rate of tuberculosis (Comparative matched analysis set): number analyzed (Participants) | 28 | 56
  Incidence rate of tuberculosis (Comparative matched analysis set) | 0.00 | 0.02
Statistical Analysis 1: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set Note: Hazard ratio, risk ratio, and risk difference for the Comparative analysis set (IPTW weighted) and for the Comparative matched analysis set could not be calculated. Also, crude hazard ratio and crude risk ratio could not be calculated; Test type: Other — Estimation; Risk Difference (RD) = 0.00, 95% CI 2-sided [-0.01 to 0.00] — Crude Risk Difference (Exposed-Reference), where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade

3. Secondary Outcome: Incidence Rate of Serious Blood Disorder
Description: The observation of serious blood disorder was expected to occur in an acute time period following any exposure. An incident event occurring during the 60-day risk window was counted in the numerator for the analysis and the person-time accrued until the first occurrence of an event, the end of the 60-day risk window, date of switch treatment, death, or the end of study period. Additionally, two types of analyses based on propensity score were conducted.
  For the full analysis set, 1 and 15 events occurred with a total of 163.5 and 2913.5 person-years in the Infliximab-Pfizer Biosimilar group and Remicade group, respectively. For the comparative analysis set, 1 and 15 events occurred with a total of 27.5 and 2913.5 person-years. For the comparative analysis set (IPTW weighted), 0.1 and 14.9 events occurred with a total of 10.4 and 2899.6 person-years. For the comparative matched analysis set, 1 and 0 events occurred with a total of 27.5 and 52.5 person-years.
Time Frame: From index date up to 60 days after last dose
Population: For the analysis of each outcome event, those patients experiencing the same outcome event during the 90-day look-back period prior to the index date were excluded. For serious blood disorder, this resulted in Full analysis set (Infliximab-Pfizer Biosimilar, n=92; Remicade, n=2093), Comparative analysis set (Infliximab-Pfizer Biosimilar, n=28; Remicade, n=2093).
Measure: Number; unit: serious blood disorder per 1 person-year
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] | Remicade (Infliximab [Genetical Recombination])
Number analyzed (Participants) | 92 | 2115
serious blood disorder per 1 person-year
  Incidence rate of serious blood disorder (Full analysis set): number analyzed (Participants) | 92 | 2093
  Incidence rate of serious blood disorder (Full analysis set) | 0.01 | 0.01
  Incidence rate of serious blood disorder (Comparative analysis set): number analyzed (Participants) | 28 | 2093
  Incidence rate of serious blood disorder (Comparative analysis set) | 0.04 | 0.01
  Incidence rate of serious blood disorder (Comparative analysis set, IPTW weighted): number analyzed (Participants) | 28 | 2093
  Incidence rate of serious blood disorder (Comparative analysis set, IPTW weighted) | 0.01 | 0.01
  Incidence rate of serious blood disorder (Comparative matched analysis set): number analyzed (Participants) | 28 | 55
  Incidence rate of serious blood disorder (Comparative matched analysis set) | 0.04 | 0.00
Statistical Analysis 1: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set, IPTW weighted; Test type: Other — Estimation; Cox Proportional Hazard = 1.22, 95% CI 2-sided [0.12 to 12.49] — Hazard Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 2: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set, IPTW weighted; Test type: Other — Estimation; Risk Ratio (RR) = 1.41, 95% CI 2-sided [0.12 to 17.14] — Risk Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 3: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set, IPTW weighted; Test type: Other — Estimation; Risk Difference (RD) = 0.00, 95% CI 2-sided [-0.05 to 0.01] — Risk Difference (Exposed-Reference), where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 4: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set Note: Hazard ratio, risk ratio, and risk difference for the comparative matched analysis set could not be calculated; Test type: Other — Estimation; Cox Proportional Hazard = 6.12, 95% CI 2-sided [0.81 to 45.94] — Crude Hazard Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 5: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set; Test type: Other — Estimation; Risk Ratio (RR) = 7.07, 95% CI 2-sided [0.93 to 53.51] — Crude Risk Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 6: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set; Test type: Other — Estimation; Risk Difference (RD) = 0.03, 95% CI 2-sided [-0.04 to 0.10] — Crude Risk Difference (Exposed-Reference), where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade

4. Secondary Outcome: Incidence Rate of Interstitial Pneumonia
Description: The observation of interstitial pneumonia was expected to occur in an acute time period following any exposure. An incident event occurring during the 60-day risk window was counted in the numerator for the analysis and the person-time accrued until the first occurrence of an event, the end of the 60-day risk window, date of switch treatment, death, or the end of study period. Additionally, two types of analyses based on propensity score were conducted.
  For the full analysis set, 5 and 42 events occurred with a total of 157.1 and 2918.8 person-years in the Infliximab-Pfizer Biosimilar group and Remicade group, respectively. For the comparative analysis set, 1 and 42 events occurred with a total of 26.2 and 2918.8 person-years. For the comparative analysis set (IPTW weighted), 0.3 and 42.1 events occurred with a total of 10.1 and 2905.0 person-years. For the comparative matched analysis set, 1 and 1 event occurred with a total of 26.2 and 52.5 person-years.
Time Frame: From index date up to 60 days after last dose
Population: For the analysis of each outcome event, those patients experiencing the same outcome event during the 90-day look-back period prior to the index date were excluded. For interstitial pneumonia, this resulted in Full analysis set (Infliximab-Pfizer Biosimilar, n=91; Remicade, n=2092), Comparative analysis set (Infliximab-Pfizer Biosimilar, n=27; Remicade, n=2092).
Measure: Number; unit: interstitial pneumonia per 1 person-year
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] | Remicade (Infliximab [Genetical Recombination])
Number analyzed (Participants) | 92 | 2115
interstitial pneumonia per 1 person-year
  Incidence rate of interstitial pneumonia (Full analysis set): number analyzed (Participants) | 91 | 2092
  Incidence rate of interstitial pneumonia (Full analysis set) | 0.03 | 0.01
  Incidence rate of interstitial pneumonia (Comparative analysis set): number analyzed (Participants) | 27 | 2092
  Incidence rate of interstitial pneumonia (Comparative analysis set) | 0.04 | 0.01
  Incidence rate of interstitial pneumonia (Comparative analysis set, IPTW weighted): number analyzed (Participants) | 27 | 2092
  Incidence rate of interstitial pneumonia (Comparative analysis set, IPTW weighted) | 0.03 | 0.01
  Incidence rate of interstitial pneumonia (Comparative matched analysis set): number analyzed (Participants) | 27 | 56
  Incidence rate of interstitial pneumonia (Comparative matched analysis set) | 0.04 | 0.02
Statistical Analysis 1: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set, IPTW weighted; Test type: Other — Estimation; Cox Proportional Hazard = 1.70, 95% CI 2-sided [0.16 to 17.61] — Hazard Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 2: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set, IPTW weighted; Test type: Other — Estimation; Risk Ratio (RR) = 1.85, 95% CI 2-sided [0.17 to 19.79] — Risk Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 3: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set, IPTW weighted; Test type: Other — Estimation; Risk Difference (RD) = 0.01, 95% CI 2-sided [-0.12 to 0.03] — Risk Difference (Exposed-Reference), where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 4: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative matched analysis set; Test type: Other — Estimation; Cox Proportional Hazard = 2.61, 95% CI 2-sided [0.15 to 45.68] — Hazard Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 5: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative matched analysis set; Test type: Other — Estimation; Risk Ratio (RR) = 2.01, 95% CI 2-sided [0.12 to 34.94] — Risk Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 6: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative matched analysis set; Test type: Other — Estimation; Risk Difference (RD) = 0.02, 95% CI 2-sided [-0.10 to 0.26] — Risk Difference (Exposed-Reference), where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 7: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set; Test type: Other — Estimation; Cox Proportional Hazard = 2.70, 95% CI 2-sided [0.37 to 19.93] — Crude Hazard Ratio Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 8: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set; Test type: Other — Estimation; Risk Ratio (RR) = 2.66, 95% CI 2-sided [0.37 to 19.31] — Crude Risk Ratio Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 9: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set; Test type: Other — Estimation; Risk Difference (RD) = 0.02, 95% CI 2-sided [-0.05 to 0.10] — Crude Risk Difference (Exposed-Reference), where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade

5. Secondary Outcome: Incidence Rate of Malignancy
Description: This study analyzed malignancy by extending follow-up time until the first incident event, death, end of the study period, or loss to follow-up. The primary analysis utilized an ever-exposed approach whereby a person always was considered exposed to the initial treatment. All malignancies were reported in the primary analysis even those that occur after the day of initial treatment. Additionally, two types of analyses based on propensity score were conducted.
  For the full analysis set, 7 and 77 events occurred with a total of 172.5 and 4480.2 person-years in the Infliximab-Pfizer Biosimilar group and Remicade group, respectively. For the comparative analysis set, 1 and 77 events occurred with a total of 27.7 and 4480.2 person-years. For the comparative analysis set (IPTW weighted), 0.0 and 76.7 events occurred with a total of 10.5 and 4458.5 person-years. For the comparative matched analysis set, 1 and 4 events occurred with a total of 27.7 and 78.4 person-years.
Time Frame: From index date up to the first incident event, death, end of the study period, or loss to follow-up
Population: For the analysis of each outcome event, those patients experiencing the same outcome event during the 90-day look-back period prior to the index date were excluded. For malignancy, this resulted in Full analysis set (Infliximab-Pfizer Biosimilar, n=89; Remicade, n=2094), Comparative analysis set (Infliximab-Pfizer Biosimilar, n=26; Remicade, n=2094).
Measure: Number; unit: malignancy per 1 person-year
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] | Remicade (Infliximab [Genetical Recombination])
Number analyzed (Participants) | 92 | 2115
malignancy per 1 person-year
  Incidence rate of malignancy (Full analysis set): number analyzed (Participants) | 89 | 2094
  Incidence rate of malignancy (Full analysis set) | 0.04 | 0.02
  Incidence rate of malignancy (Comparative analysis set): number analyzed (Participants) | 26 | 2094
  Incidence rate of malignancy (Comparative analysis set) | 0.04 | 0.02
  Incidence rate of malignancy (Comparative analysis set, IPTW weighted): number analyzed (Participants) | 26 | 2094
  Incidence rate of malignancy (Comparative analysis set, IPTW weighted) | 0.00 | 0.02
  Incidence rate of malignancy (Comparative matched analysis set): number analyzed (Participants) | 26 | 56
  Incidence rate of malignancy (Comparative matched analysis set) | 0.04 | 0.05
Statistical Analysis 1: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set, IPTW weighted; Test type: Other — Estimation; Cox Proportional Hazard = 0.18, 95% CI 2-sided [0.02 to 1.85] — Hazard Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 2: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set, IPTW weighted; Test type: Other — Estimation; Risk Ratio (RR) = 0.19, 95% CI 2-sided [0.02 to 1.99] — Risk Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 3: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set, IPTW weighted; Test type: Other — Estimation; Risk Difference (RD) = -0.01, 95% CI 2-sided [-0.17 to 0.00] — Risk Difference (Exposed-Reference), where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 4: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative matched analysis set; Test type: Other — Estimation; Cox Proportional Hazard = 0.63, 95% CI 2-sided [0.07 to 6.00] — Hazard Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 5: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative matched analysis set; Test type: Other — Estimation; Risk Ratio (RR) = 0.71, 95% CI 2-sided [0.08 to 6.61] — Risk Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 6: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative matched analysis set; Test type: Other — Estimation; Risk Difference (RD) = -0.01, 95% CI 2-sided [-0.10 to 0.21] — Risk Difference (Exposed-Reference), where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 7: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set; Test type: Other — Estimation; Cox Proportional Hazard = 2.07, 95% CI 2-sided [0.28 to 15.22] — Crude Hazard Ratio Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 8: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set; Test type: Other — Estimation; Risk Ratio (RR) = 2.10, 95% CI 2-sided [0.29 to 15.08] — Crude Risk Ratio of Exposed/Reference, where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade
Statistical Analysis 9: Comparison: Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] vs Remicade (Infliximab [Genetical Recombination]); Comparative analysis set; Test type: Other — Estimation; Risk Difference (RD) = 0.02, 95% CI 2-sided [-0.05 to 0.09] — Crude Risk Difference (Exposed-Reference), where Exposed is Infliximab-Pfizer Biosimilar and Reference is Remicade

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not planned to be collected during the study.
Description: Minimum criteria for reporting an adverse event (i.e., identifiable patients, identifiable reporter, a suspect product, and event) could not be met. Hence, adverse events were not collected or reported.
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar3] | Remicade (Infliximab [Genetical Recombination])
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT05796245/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT05796245/SAP_001.pdf